CLINICAL TRIAL: NCT01431547
Title: A Phase I Study of Monotherapy Dalotuzumab and Ridaforolimus-Dalotuzumab Combination Treatment in Pediatric Patients With Advanced Solid Tumors
Brief Title: Study of Dalotuzumab Alone and With Ridaforolimus in Pediatric Participants With Advanced Solid Tumors (MK-8669-062 AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-062
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — dalotuzumab; ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Dalotuzumab (Experimental)
  Interventions: Drug: dalotuzumab
- Parts 2 and 3: Dalotuzumab + ridaforolimus (Experimental)
  Interventions: Drug: dalotuzumab; Drug: ridaforolimus

INTERVENTIONS:
Drug: dalotuzumab — For Part 1: dalotuzumab, intravenously (IV) over 60 minutes every three weeks, dose based on participant body surface area (BSA), starting dose of 900 mg/m^2, and escalated for successive cohorts of participants until MTD is found
  Arms: Part 1: Dalotuzumab
Drug: dalotuzumab — For Part 2: dalotuzumab IV over 60 minutes every three weeks, dose based on participant BSA, starting at the lowest tolerated dose that met PK target levels in Part 1. For Part 3: dalotuzumab IV over 60 minutes every three weeks, dose based on participant BSA, at the dose level identified for combination therapy in Part 2
  Arms: Parts 2 and 3: Dalotuzumab + ridaforolimus
Drug: ridaforolimus — For Part 2: ridaforolimus 10 mg enteric coated tablets, orally, on 5 consecutive days each week, dose based on participant BSA, at 1 dose level lower than the MTD or highest dose level used in the companion study MK-8669-056. For Part 3:ridaforolimus 10 mg enteric coated tablets, orally, on 5 consecutive days each week, dose based on participant BSA, at the dose level identified for combination therapy in Part 2
  Other Names: MK-8669
  Arms: Parts 2 and 3: Dalotuzumab + ridaforolimus

SUMMARY:
This is a study of dalotuzumab given as monotherapy and in combination with ridaforolimus for pediatric participants with advanced solid tumors. This study will have three parts. Part 1 will find a maximum tolerated dose (MTD) and collect pharmacokinetic (PK) data for dalotuzumab alone. Part 2 will find an MTD and collect PK data for dalotuzumab in combination with ridaforolimus. Part 3 will be an expansion cohort at the recommended Phase 2 dose (RPTD) found in Part 2 to confirm the RPTD and look at the potential efficacy of the combination therapy.

ELIGIBILITY:
Inclusion criteria:

* Participants of age 3 to 17 years for Part 1 of the study and age 6 to 17 years for Parts 2 and 3 of the study
* Histologic or cytologic diagnosis of a malignant solid tumor, including tumors of the central nervous system and lymphoma, that have progressed despite standard therapy or for which no effective standard therapy is known.
* Measurable or non-measurable disease for Parts 1 and 2; measurable disease for Part 3
* Parts 2 and 3: must be able to swallow tablets
* Performance Status: Lansky Play Scale ≥70 for children <10 years of age; Karnofsky score ≥70 for children ≥10 to <16 years; or Eastern Cooperative Oncology Group (ECOG) Status 0-2 for patients age 16 and older
* Adequate organ function
* For females of reproductive potential, a negative pregnancy test must be documented within 72 hours of receiving the first dose of study medication
* Participants of reproductive potential must agree to use (or have their partner use) adequate contraception throughout the study, starting with Visit 1 through 30 days after the last dose of study drug

Exclusion criteria:

* Currently receiving any other investigational agents or using any investigational devices
* Leukemia
* Previously received dalotuzumab or other IGF-1R inhibitors for Part 1
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dalotuzumab or ridaforolimus
* Persistent acute toxicity from previous therapy ≥Grade 2 (excluding alopecia, neuropathy, or hearing loss)
* Uncontrolled intercurrent illness despite adequate therapy
* Pregnant or breastfeeding
* For Parts 2 and 3: requirement for concurrent treatment with medications that are inducers or inhibitors of cytochrome P450 (CYP3A)
* Poorly controlled Type 1 or 2 diabetes

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) while receiving dalotuzumab alone | First 21 days of treatment
Number of participants with DLTs while receiving dalotuzumab and ridaforolimus combination therapy | First 21 days of treatment
Dalotuzumab mean serum trough concentration | Day 22, pre-dose (Part 1)
Dalotuzumab mean serum trough concentration in combination therapy | Day 22, pre-dose (Part 2)
Ridaforolimus geometric mean area under the concentration curve from Hour 0 to Hour 24 (AUC [0-24]) in combination therapy | Cycle 1, Day 5 (Part 2)

REFERENCES:
- [Result] Frappaz D, Federico SM, Pearson AD, Gore L, Macy ME, DuBois SG, Aerts I, Iannone R, Geschwindt R, Van Schanke A, Wang R, Geoerger B. Phase 1 study of dalotuzumab monotherapy and ridaforolimus-dalotuzumab combination therapy in paediatric patients with advanced solid tumours. Eur J Cancer. 2016 Jul;62:9-17. doi: 10.1016/j.ejca.2016.03.084. Epub 2016 May 10. PMID 27185573